CLINICAL TRIAL: NCT07223892
Title: A Prospective Controlled Trial Evaluating the Efficacy of Carbonlife Amniotic Tissue Product in the Treatment of Chronic Wounds: A Stratified Analysis by Wound Etiology and Care Setting
Brief Title: Efficacy of Carbonlife Amniotic Tissue Product in the Treatment of Chronic Wounds
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bardia Anvar (Industry)
Collaborators: Carbon Life Sciences (Industry)
Responsible Party: Sponsor-Investigator, Bardia Anvar, Principle Investigator, Carbon Life Sciences
Organization: Carbon Life Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Carbonlife
Record Dates: First submitted 2025-10-23; First posted 2025-11-03 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Chronic Wounds; Venous Leg Ulcers (VLUs); Diabetic Foot Ulcers (DFUs); Arterial Ulcers; Pressure Ulcers; Burn Wounds; Trauma Wounds; Surgical Wounds
Keywords: chronic wounds
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer; Burns; Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATP Treatment Group (Experimental): Application of Carbonlife ATP per manufacturer's instructions along with standard wound care.
  Interventions: Biological: Amniotic Tissue Allograft
- Standard Wound Care Group (No Intervention): Patients will not received Amnionic Tissue Product to treat chronic wounds. Participants will receive:
  * Wound debridement as needed
  * Dressing selection based on wound characteristics
  * Compression therapy for venous ulcers (if indicated)
  * Offloading for pressure ulcers (if indicated)

INTERVENTIONS:
Biological: Amniotic Tissue Allograft — The amniotic tissue products will be used to treat patients with chronic wounds to determine if a higher incidence of wound closure or reduction in devitalized tissue occurs.
  Other Names: Amniotic Tissue Graft; Amniotic Tissue Product
  Arms: ATP Treatment Group

SUMMARY:
Chronic wounds constitute a significant global health burden, affecting millions of individuals and contributing to increased morbidity, diminished quality of life, and rising healthcare costs. These wounds are characterized by delayed healing and are often associated with complex etiologies and prolonged treatment courses. This study aims to evaluate the clinical efficacy and cost-effectiveness of Carbonlife amniotic tissue products (ATPs) compared to standard wound care in the management of chronic wounds. A prospective, controlled clinical trial will be conducted across diverse care settings and patient populations with varying wound etiologies. Participants will be stratified by wound type and treatment environment to enable subgroup analyses. The primary endpoint will assess wound healing outcomes, while secondary endpoints will include quality-of-life measures and healthcare resource utilization. The study is designed to generate high-quality evidence regarding the therapeutic value of ATPs in chronic wound management. Stratified analyses will provide insights into the differential effectiveness of ATPs across clinical contexts. Findings are anticipated to have implications for clinical practice guidelines and healthcare policy, with the goal of improving patient outcomes and optimizing resource allocation in wound care.

ELIGIBILITY:
Inclusion Criteria:

* Facilities and centers with the capacity to follow strict treatment and care guidelines for patients.
* Adults aged 18 years or older.
* Presence of a chronic wound (defined as a wound that has not shown significant improvement in 4 weeks) of any of the following etiologies: Diabetic foot ulcers, Venous leg ulcers, Arterial ulcers, Pressure ulcers, Burns, Trauma, Surgical
* Wound size greater than 1 cm²
* Ability to provide informed consent

Exclusion Criteria:

* Presence of active osteomyelitis
* Untreated malignancy in the wound area
* Known allergy to components of ATPs
* Pregnant or breastfeeding women
* Patients receiving immunosuppressive therapy
* Patients with a life expectancy of less than 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | 12 Weeks
  Complete wound closure, defined as 100% epithelialization without drainage.

SECONDARY OUTCOMES:
Duration of Wound Closure | This is dependent on the time the wound closes, 12 - 20 week estimate.
  The time it takes to close the wound.
Wound Area Reduction | 12 Weeks
  Percentage of wound area reduction at 4, 8, and 12 weeks.
Adverse Events | 12 Weeks
  Tracking the number of adverse events.
Numerical Pain Assessment | 12 Weeks
  Using the Numerical Pain Assessment, patients will rate their level of pain on a scale from 1 to 10 (1 being no pain and 10 being excruciating pain).
Visual Analogue Pain Assessment | 12 Weeks
  Using the Visual Analogue Pain Assessment, patients unable to rate their pain numerically, will choose the face that best represents their level of pain. Their response will be scored based on the number (1 through 10) associated with that face. 1 represents no pain, and 10 represents excruciating pain.

IPD SHARING:
Plan to Share IPD: Yes
The specific IPD that may be included in the reports and publications stemming from this clinical study may include, but is not limited to: age, gender, details on wound etiologies and diagnostics, responses to pain assessments, adverse event reports, comprehensive treatment details, and clinical therapy outcomes. All shared data would be de-identified and used per patient authorization.